CLINICAL TRIAL: NCT06334120
Title: Post-marketing Surveillance Study for Approved Darolutamide Use in Korean Patients
Brief Title: An Observational Study to Learn More About the Safety of Darolutamide in Men With Prostate Cancer in Korea
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20654
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-metastatic Castration-resistant Prostate Cancer; Metastatic Hormone-sensitive Prostate Cancer
MeSH Terms: interventions — darolutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male patients with nmCRPC or mHSPC: Male patients with a diagnosis of non-metastatic castration-resistant prostate cancer (nmCRPC) or metastatic hormone-sensitive prostate cancer (mHSPC) will be enrolled after the decision for treatment with Darolutamide has been made by the investigator.
  Interventions: Drug: Darolutamide (Nubeqa, BAY1841788)

INTERVENTIONS:
Drug: Darolutamide (Nubeqa, BAY1841788) — The decision on the dose and duration of treatment is solely at the discretion of the treating physician, based on the recommendations written in the local product information.

SUMMARY:
This is an observational study in which participants receive a treatment which is already available for doctors to prescribe for non-metastatic castration-resistant prostate cancer (nmCRPC) or metastatic hormone-sensitive prostate cancer (mHSPC). nmCRPC is a prostate cancer that has not yet spread to other parts of the body and does not respond to lowering testosterone in the body. mHSPC is a prostate cancer that has spread to other parts of the body and can be treated by lowering testosterone levels.

This study looks at the safety of the study drug, darolutamide, in Korean patients with nmCRPC or mHSPC. Darolutamide is currently available for doctors to prescribe to men with nmCRPC or mHSPC. It works by attaching to the special molecules called androgen receptors (AR) within prostate cells and blocks hormones called androgens from attaching to AR, which helps delay cancer growth.

To learn more about the safety of Darolutamide, the researchers will study whether the participants have adverse events. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments. The researchers will also learn more about how well darolutamide is working in these participants.

During this study, the researchers will collect information from the medical records of patients who have been prescribed darolutamide by their doctors.

Each participant will be in this study for 1 year. The whole study will last about 6 years. During this time, the participants will visit their doctor every 2 to 4 months as part of their usual care. At these visits, the doctors will do scans to check the patients' cancer and take blood samples. The patients will answer questions about any medications they are taking and whether they have any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male aged ≥19 years
* Patients with high risk nmCPRC

  * Castrate level of serum testosterone (< 1.7 nmol/l [50 ng/dL])
  * PSA doubling time < 10 months
* Patients with mHSPC

  * histologically or cytologically confirmed prostate cancer, and metastases detected on bone scanning, contrast-enhanced computed tomography (CT), or magnetic resonance imaging (MRI).
  * be candidates for androgen-deprivation therapy with/without docetaxel.
* Patients for whom the decision to initiate treatment with Darolutamide as a first time was made as per investigator's routine treatment practice
* Written informed consent from subject or legal representative; assent from subject when appropriate

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice
* Participants with contraindication according to the locally approved prescribing information

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been prescribed Darolutamide for a medically appropriate use will be eligible to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number, severity of adverse events (including SAEs) | From the date that the patient signed the informed consent to 30 days after the end of the treatment (up to 52 weeks)
  SAE stands for serious adverse event. An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number, severity of adverse drug reactions (including SADRs) | From the date that the patient signed the informed consent to 30 days after the end of the treatment (up to 52 weeks)
  SADR stands for serious adverse drug reaction. An ADR is any AE judged by investigator as having a reasonable suspected causal relationship to Darolutamide.
The outcome of (serious) adverse events | From the date that the patient signed the informed consent to 30 days after the end of the treatment (up to 52 weeks)
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
The outcome of (serious) adverse drug reactions | From the date that the patient signed the informed consent to 30 days after the end of the treatment (up to 52 weeks)
  An ADR is any AE judged by investigator as having a reasonable suspected causal relationship to Darolutamide.

SECONDARY OUTCOMES:
Metastasis-free survival (MFS) by nmCRPC indication | Up to 52 weeks
  MFS is defined as the time (months) from the initiation of Darolutamide treatment to the date of first observed metastasis.
Time to first symptomatic skeletal event (SSE) by nmCRPC indication | Up to 52 weeks
  Time to SSE is defined as the time (months) from the initiation of Darolutamide treatment to the date of first diagnosed skeletal-related event.
Time to prostate-specific antigen (PSA) progression by nmCRPC indication | Up to 52 weeks
  Time to PSA progression is defined as the time (months) from the initiation of Darolutamide treatment to the date at which PSA is recorded at ≥25% increase above the nadir (lowest screening or baseline) value along with an increase in absolute value of ≥2 ng/mL above nadir.
Overall survival by nmCRPC indication | Up to 52 weeks
  Overall survival is defined as the time (months) from the initiation of Darolutamide treatment until death from any cause.
Time to Castration-Resistant Prostate Cancer (CRPC) by mHSPC indication | Up to 52 weeks
  Time to mCRPC, defined as the time to PSA progression with serum testosterone being at castrate level <0.50 ng/mL, or the time to progression by soft tissue/visceral lesions or time to progression by bone lesions, whatever comes first.
Time to first symptomatic skeletal event (SSE) by mHSPC indication | Up to 52 weeks
  Time to SSE is defined as the time (months) from the initiation of Darolutamide treatment to the date of first diagnosed skeletal-related event.
Time to prostate-specific antigen (PSA) progression by mHSPC indication | Up to 52 weeks
  Time to PSA progression is defined as the time (months) from the initiation of Darolutamide treatment to the date at which PSA is recorded at ≥25% increase above the nadir (lowest screening or baseline) value along with an increase in absolute value of ≥2 ng/mL above nadir.
Overall survival by mHSPC indication | Up to 52 weeks
  Overall survival is defined as the time (months) from the initiation of Darolutamide treatment until death from any cause.
Time to initiation of subsequent anti-cancer therapy by mHSPC indication | Up to 52 weeks
  Time to initiation of subsequent anti-cancer therapy is defined as the time (months) from the initiation of Darolutamide treatment to the date of first administration of any subsequent anti-cancer therapy after discontinuation of Darolutamide.
Radiological progression (Soft tissue/ Bone metastasis) by mHSPC indication | Up to 52 weeks
  Radiological progression is defined as the time (months) from the start of Darolutamide treatment to the date of first documentation of radiological progressive disease or death due to any cause, whichever occurs first.
Radiological Progression-Free Survival (rPFS) by mHSPC indication | Up to 52 weeks
  Radiographic Progression-Free Survival (rPFS) is defined as the time (months) from the initiation of Darolutamide treatment to the date of the first radiologically confirmed disease progression or death from any cause, whichever occurs first.
Duration of Darolutamide treatment | Up to 52 weeks
  Duration of Darolutamide treatment is defined as the time (months) from the start of Darolutamide treatment to the day of permanent discontinuation of Darolutamide (including death).
Reasons for ending Darolutamide | Up to 52 weeks
Dosage and dose modification of Darolutamide | Up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple locations, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.